CLINICAL TRIAL: NCT00674440
Title: Localization of Focal Forms of Hyperinsulinism of Infancy With 18F-labeled L-fluoro-DOPA PET Scan
Brief Title: Utility of [F-18] fluoroDOPA for Neonatal Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa States, Attending Physician/Radiologist, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-003683; FD-R-003457-01 (Other Grant/Funding Number: FDA orphan drug grant)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Congenital Hyperinsulinism; Hyperinsulinism; Persistent Hyperinsulinemic Hypoglycemia of Infancy; CHI; PHHI
Keywords: Congenital Hyperinsulinism; Hyperinsulinism; Persistent Hyperinsulinemic Hypoglycemia of Infancy; CHI; PHHI; F-DOPA; L-fluoro-dihydroxyphenylalanine
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects who had PET and surgery (Experimental): Children diagnosed with hyperinsulinism who have failed other non-surgical interventions and are candidates to be scheduled for surgery for partial pancreatectomy. Eligible children will undergo PET imaging with F-DOPA prior to surgery.
  Interventions: Drug: F-DOPA; Radiation: PET scan

INTERVENTIONS:
Drug: F-DOPA — 0.08-0.16 mCi/kg once
  Other Names: 18F-labeled L-fluorodeoxyphenylalanine; 18F-DOPA
Radiation: PET scan

SUMMARY:
Children with congenital hyperinsulinism (CHI) have low blood sugar, and some of these children may require surgery. In this study, researchers affiliated with the University of Pennsylvania will test how well a radioactive drug (called F-DOPA) can detect a form of hyperinsulinism that may be cured by surgery. Eligible participants in this study will have positron emission tomography (PET) scans with F-DOPA prior to surgery.

DETAILED DESCRIPTION:
For children with congenital hyperinsulinism (CHI), low blood sugar is caused by cells in the pancreas that release too much insulin. Some children with CHI have these cells throughout their pancreas; others have them located in specific areas of the pancreas. Children who have them located in specific areas of the pancreas may be cured with surgery. F-DOPA is a radioactive drug that may go to these very cells. F-DOPA can also be used for positron emission tomography (or PET), an imaging technique used in nuclear medicine departments. In this study, researchers will test the possibility of using PET with F-DOPA in the diagnosis of children with hyperinsulinism.

ELIGIBILITY:
Inclusion Criteria:

* Any age, but primarily infants 0-6 months.
* Children with confirmed diagnosis of congenital hyperinsulinism.

Exclusion Criteria:

* Cases in which surgery will not be considered by parents or guardians.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J States, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hardy OT, Litman RS. Congenital hyperinsulinism - a review of the disorder and a discussion of the anesthesia management. Paediatr Anaesth. 2007 Jul;17(7):616-21. doi: 10.1111/j.1460-9592.2007.02192.x. PMID 17564642
- [Background] Otonkoski T, Nanto-Salonen K, Seppanen M, Veijola R, Huopio H, Hussain K, Tapanainen P, Eskola O, Parkkola R, Ekstrom K, Guiot Y, Rahier J, Laakso M, Rintala R, Nuutila P, Minn H. Noninvasive diagnosis of focal hyperinsulinism of infancy with [18F]-DOPA positron emission tomography. Diabetes. 2006 Jan;55(1):13-8. PMID 16380471
- [Background] Ribeiro MJ, Boddaert N, Delzescaux T, Valayannopoulos V, Bellanne-Chantelot C, Jaubert F, Verkarre V, Nihoul-Fekete C, Brunelle F, Lonlay P. Functional imaging of the pancreas: the role of [18F]fluoro-L-DOPA PET in the diagnosis of hyperinsulinism of infancy. Endocr Dev. 2007;12:55-66. doi: 10.1159/000109605. PMID 17923769
- [Background] Subramaniam RM, Karantanis D, Peller PJ. [18F]Fluoro-L-dopa PET/CT in congenital hyperinsulinism. J Comput Assist Tomogr. 2007 Sep-Oct;31(5):770-2. doi: 10.1097/RCT.0b013e318031f55c. PMID 17895790
- [Background] Ribeiro MJ, Boddaert N, Bellanne-Chantelot C, Bourgeois S, Valayannopoulos V, Delzescaux T, Jaubert F, Nihoul-Fekete C, Brunelle F, De Lonlay P. The added value of [18F]fluoro-L-DOPA PET in the diagnosis of hyperinsulinism of infancy: a retrospective study involving 49 children. Eur J Nucl Med Mol Imaging. 2007 Dec;34(12):2120-8. doi: 10.1007/s00259-007-0498-y. Epub 2007 Jul 28. PMID 17661030
- [Background] de Lonlay P, Simon-Carre A, Ribeiro MJ, Boddaert N, Giurgea I, Laborde K, Bellanne-Chantelot C, Verkarre V, Polak M, Rahier J, Syrota A, Seidenwurm D, Nihoul-Fekete C, Robert JJ, Brunelle F, Jaubert F. Congenital hyperinsulinism: pancreatic [18F]fluoro-L-dihydroxyphenylalanine (DOPA) positron emission tomography and immunohistochemistry study of DOPA decarboxylase and insulin secretion. J Clin Endocrinol Metab. 2006 Mar;91(3):933-40. doi: 10.1210/jc.2005-1713. Epub 2006 Jan 10. PMID 16403819
- [Result] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Scheuermann JS, Ernst LM, Freifelder R, Zhuang H, MacMullen C, Becker S, Adzick NS, Divgi C, Alavi A, Stanley CA. Accuracy of [18F]fluorodopa positron emission tomography for diagnosing and localizing focal congenital hyperinsulinism. J Clin Endocrinol Metab. 2007 Dec;92(12):4706-11. doi: 10.1210/jc.2007-1637. Epub 2007 Sep 25. PMID 17895314
- [Result] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Suchi M, Ruchelli E, Zhuang H, Ganguly A, Freifelder R, Adzick NS, Alavi A, Stanley CA. Diagnosis and localization of focal congenital hyperinsulinism by 18F-fluorodopa PET scan. J Pediatr. 2007 Feb;150(2):140-5. doi: 10.1016/j.jpeds.2006.08.028. PMID 17236890
- See also: The Congenital Hyperinsulinism Center at The Children's Hospital of Philadelphia — http://hyperinsulinism.chop.edu.
- See also: International non-profit organization created by parents/families based in the United States — http://www.congenitalhi.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2004 to December 2008, the study team recruited and enrolled 106 subjects referred to the Congenital Hyperinsulinism Center at the Children's Hospital of Philadelphia who were potential candidates for partial pancreatectomy surgery if focal lesions were suspected and were able to be localized.
Pre-assignment Details: The participants newly diagnosed with hypersulinism required surgery for hyperinsulinism. A subset of patients who seemed to respond to medical therapy or had continued hyperinsulinism after surgery were also included. All subjects were consented for PET scan and were eligible for surgery. 105 patients underwent F-DOPA PET with the same research procedures.
Groups:
- All Subjects Consented: There were 106 subjects consented to participate. 105 actually underwent PET scan.
Period: Overall Study
Arm/Group | All Subjects Consented
Started | 106
Completed | 95 (Subjects who had PET and surgery and were evaluable)
Not Completed | 11
Not completed — consented but not scanned (Withdrawn due to genetics) | 1
Not completed — did not have surgery, so unevaluable | 7
Not completed — had atypical histology or had second PET scan after initial surgery - not counted twice | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Who Consented: These demographics include all subject recruited who consented whether they are evaluable or not
Arm/Group | Subjects Who Consented
Number analyzed (Participants) | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 106
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 73
  More than one race | 23
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94
  Canada | 7
  Israel | 1
  Brazil | 1
  Curacao | 1
  Iran | 1
  Saudi Arabia | 1

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy of FDOPA PET to Identify Focal Forms of Hyperinsulinism
Description: Comparison of PET scan results with outcome of surgery and histopathology results confirmed as focal or diffuse
Time Frame: up to 1 month post surgical intervention
Population: An F-DOPA PET/CT imaging study was performed and reported prior to surgery. This data includes surgical histopathology confirmed as focal or diffuse. 95 of the 106 original consented participants had surgical results that were evaluable. (1 consented but never scanned, 7 did not have surgery, 3 had surgery but were excluded for atypical histology that did not fit classic focal or diffuse or had second PET scan after initial surgery therefore not counted twice).
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Who Had PET and Surgery: To determine the sensitivity and specificity of 18F-DOPA PET/CT for the detection of a focal pancreatic lesion in infants and children with poorly controlled hyperinsulinemic hypoglycemia.
Arm/Group | Subjects Who Had PET and Surgery
Number analyzed (Participants) | 95
Participants
  True Negatives (PET diffuse/surgery diffuse) | 40
  False negatives (PET diffuse/surgery focal): | 6
  False positives (PET focal/surgery diffuse): | 3
  True positives (PET focal/surgery focal): | 46
Statistical Analysis 1: Comparison: Subjects Who Had PET and Surgery; Test type: Other; Sensitivity = 93.0, 95% CI 2-sided [80.9 to 98.5]
Statistical Analysis 2: Comparison: Subjects Who Had PET and Surgery; Test type: Other; Specifity = 88.5, 95% CI 2-sided [76.6 to 95.6]

2. Secondary Outcome: Safety of F-DOPA PET
Description: Number of Participants with Adverse Events
Time Frame: 72 hours maximum or prior to pancreatic surgery
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Who Had PET: This group included the 105 subjects who had F-DOPA PET scan whether they had surgery or not
Arm/Group | All Subjects Who Had PET
Number analyzed (Participants) | 105
Participants | 0

ADVERSE EVENTS:
Time Frame: Reviewed within 72 hours post PET or prior to pancreatic surgery (which ever was first).
Description: Included all participants who had PET(whether or not they also had surgery).
Groups:
- All Subjects Who Had PET: Obtain safety and efficacy data on the use of 18-labeled L-fluorodeoxyphenylalanine (18F-DOPA) PET imaging in children with HI for the clinical indication of localizing a focal lesion
  18 F-DOPA: 1 time injection of 0.08 - 0.16 mCi/kg of 18F-DOPA
Arm/Group | All Subjects Who Had PET
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 0/105

LIMITATIONS AND CAVEATS:
Some subjects have atypical disease that is neither focal or diffuse. Rapid genetic test results were not available at the beginning of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes